CLINICAL TRIAL: NCT04825990
Title: Pembrolizumab and Olaparib in Recurrent/Metastatic, Platinum Resistant Nasopharyngeal Cancer
Acronym: POINT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POINT
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — pembrolizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Treatment (Experimental): Patients will receive pembrolizumab 200 mg intravenously (IV) on Day 1 of every 3-week dosing cycle (Q3W) and olaparib 300 mg capsules twice a day (BID) every day starting from Day 1 of Cycle 1. Treatment with protocol therapy will continue until objective disease progression, any prohibitive toxicity or until a maximum of 35 treatment cycles (up to 2 years).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg pembrolizumab every 3 weeks plus 300 mg olaparib twice a day (BID) every day starting from Day 1 of Cycle 1.
  Other Names: olaparib

SUMMARY:
Recurrence rate after curative treatment for locally advanced Nasopharyngeal carcinoma (NPC) is reported varying from 15% to 30% of cases, while approximately 5-11% of patients present with de novo metastatic disease.

In NPC, the immunogenicity of the cancer cell is derived from accumulated somatic mutations, but also from genomic and proteomic differences between host and Epstein Barr Virus (EBV). However, anti-cancer immune response tends to be feeble. This impaired anti-cancer immunity could be attributed to multiple factors including strategies to escape anti-cancer immunity. One of this is switch to immunosuppressive microenvironment, as well as aberrant negative co-stimulatory signals like PD-L1, that is over expressed in NPC. In 2017, the landmark KEYNOTE-028 trial firstly reported promising antitumor activities and safety profiles of pembrolizumab in previously treated RM-NPC Overall, after the treatment of PD-1 inhibitors, about 25% and 60% of the recurrent or metastatic nasopharyngeal carcinoma patients achieved ORR and DCR, respectively, with a profile of toxicities in line with the use of immune checkpoint inhibitors in other diseases.

Recently, it was found that some non-BRCA-mutated tumors often harbor other alterations in HR genes except for germline BRCA deleterious mutations, thus making these tumors could benefit from PARPi treatment.

PARP could contribute to resistance to chemotherapy induced DNA damage, NPC cell platinum resistant could use PARP to repair and escape apoptosis. In nasopharyngeal carcinoma PARP1 is overexpressed in comparison with normal nasopharyngeal cells, LMP1 (latent membrane protein one) activates PARP1 and increases Poly(ADP-ribos)ylation (PARylation) through PARP1. A preclinical study demonstrates that LMP1+ cells are more sensitive to PARP1 inhibition.

After receiving PARPi treatment, accumulated chromosome rearrangements generate plenty of neoantigens and elevate the immunogenicity of tumor, PARPi-mediated acute inflammation remodels tumor immune microenvironment and drives a systemic Th1-skewing immune response.

Patients in the POINT trial will receive pembrolizumab 200 mg intravenously (IV) on Day 1 of every 3-week dosing cycle (Q3W) and olaparib 300 mg capsules twice a day (BID) every day starting from Day 1 of Cycle 1. Treatment with protocol therapy will continue until objective disease progression, any prohibitive toxicity or until a maximum of 35 treatment cycles (up to 2 years).

DETAILED DESCRIPTION:
Before any study specific procedure is performed the patient will sign an informed consent form.

Every effort should be done to obtain a new tumor biopsy from relapsed-metastatic disease, but a new biopsy is not necessary to participate to the study.

Patients will undergo radiologic staging investigations according to guidelines, including pre-treatment head and neck MRI and whole body FDG-PET (or thorax and abdomen CT scan) and clinical evaluation with fiberendoscopy.

Patients will receive pembrolizumab 200 mg intravenously (IV) on Day 1 of every 3-week dosing cycle (Q3W) and olaparib 300 mg capsules twice a day (BID) every day starting from Day 1 of Cycle 1. Treatment with protocol therapy will continue until objective disease progression, any prohibitive toxicity or until a maximum of 35 treatment cycles (up to 2 years).

Patients who must discontinue one of the two drugs in the combination due to adverse events may continue the study with the other combination drug. Once patients have been discontinued from study treatment, other treatment options will be at the discretion of the investigator.

Dose reductions will be allowed according to protocol-specified rules. Tumor response will be evaluated by clinical/endoscopic evaluation every 3 weeks and by radiological imaging every 9 weeks (±7 days) since treatment start. After the first year, the radiological imaging frequency can be modified as clinically indicated. Radiologic response will be assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

Blood samples for plasmatic EBV-DNA analysis will be performed at baseline, and, if positive, at week 3, week 9 and then every 9 weeks since treatment start (however in concomitance with the radiological imagining) and at every follow up visit (in case of EBER-positive tumor).

Patients will be evaluated for treatment safety at each clinical visit by means of clinical and laboratory exams. All adverse events will be recorded by Common Terminology Criteria for Adverse Events (CTCAE), version 5.0; the investigator will assess whether those events are drug related or not. All enrolled patients will be included in overall safety analyses.

Change in the Quality-of-Life (QoL) since baseline using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module (EORTC QLQ-HN43) will be evaluated at first visit, every 9 weeks during treatment and at the follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years old
2. The participant (or legally acceptable representative) provides written informed consent.
3. Histologically confirmed diagnosis of nasopharyngeal carcinoma.
4. Disease not amenable of surgical resection or irradiation with curative intent.
5. Disease progressing within 6 months since previous platinum-based systemic treatment (as concomitant to RT or as first line treatment for RM NPC).
6. Male participants:

   A male participant must agree to use contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.
7. Female participants:

   A female participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 4 months after the last dose of study treatment.

   A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
   * Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   * A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 4 months after the last dose of study treatment.
8. Measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the start of study treatment.
10. Patients must have a life expectancy ≥ 16 weeks.
11. Adequate organ function as defined in the following table (Table 5.1). Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

1. WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
3. Prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy or alopecia may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Prior radiotherapy within 2 weeks of study intervention start. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
6. Currently participating in or has participated in a study with an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as the last dose of the previous investigational agent was received at least 4 weeks before enrollment
7. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.

   Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers
9. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided those are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Severe hypersensitivity (≥Grade 3) to study treatment drugs and/or any of its excipients.
11. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. History of (non-infectious) pneumonitis that required steroids or has currently pneumonitis.
13. Active infection requiring systemic therapy.
14. Known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority.
15. History of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA qualitative is detected) infection.

    Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Known history of active Bacillus Tuberculosis.
17. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
18. Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
19. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
20. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study therapy is 2 weeks.
21. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting study therapy is 5 weeks for enzalutamide or phenobarbital and 3 weeks for the other agents.
22. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
23. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
24. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
25. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2028-03-24 (Estimated)

PRIMARY OUTCOMES:
ORR | Week 27
  Objective Response Rate (ORR) as Assessed by Investigators according to Response Evaluation Criteria in Solid Tumors Version 1.1 by the 3rd radiological examination (week 27).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Asst Degli Spedali Civili Di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No